CLINICAL TRIAL: NCT02188719
Title: Donor-Alloantigen-Reactive Regulatory T Cell (darTreg) Therapy in Liver Transplantation (RTB-002)
Brief Title: Donor-Alloantigen-Reactive Regulatory T Cell (darTregs) in Liver Transplantation
Acronym: deLTa
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The trial could not be completed within the grant timeline.
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Rho Federal Systems Division, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DAIT RTB-002; R34AI095135 (NIH); U01AI110658 (NIH); NIAID CRMS ID#: 20182 (Other: DAIT NIAID)
Record Dates: First submitted 2014-07-10; First posted 2014-07-14 (Estimated); Results first posted 2020-07-20 (Actual); Last update posted 2020-09-22 (Actual); Status verified 2020-09

CONDITIONS: Liver Transplantation
Keywords: Donor-Alloantigen-Reactive Regulatory T Cell Therapy; Tregs; Cell- and Tissue-Based Therapy; Immunotherapy, Adoptive; Liver Transplantation
MeSH Terms: interventions — Antilymphocyte Serum; thymoglobulin; Everolimus; Tacrolimus; Mycophenolic Acid; Prednisone; Methylprednisolone Hemisuccinate; Acetaminophen; Diphenhydramine; Ganciclovir; Valganciclovir; Leukapheresis; Blood Specimen Collection; Phlebotomy; Liver Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Cohort 1 - Treg-supportive IS only (Experimental): 3 subjects (Cohort 1a) at site 1 (UCSF) and 3 subjects (Cohort 1b) from site 2 (Mayo Rochester) will receive Treg-Supportive immunosuppression (IS) regimen and will not receive Donor-Alloantigen-Reactive T Regulatory Cells (darTregs). Progression from one cohort to the next will depend on the cumulative incidence of sentinel adverse events.
  Interventions: Biological: Anti-Thymocyte Globulin - Rabbit; Drug: Everolimus; Drug: Tacrolimus; Drug: Mycophenolate mofetil; Drug: Prednisone; Drug: Anti-Infective Prophylaxis; Procedure: Blood draws; Procedure: Liver biopsies; Procedure: Liver transplantation
- Cohort 2 - darTreg infusion,50 million(range 25 to 60 million) (Experimental): At least 3 subjects will receive a single infusion of 50 million darTregs. Progression from one cohort to the next will depend on the cumulative incidence of sentinel adverse events.
  Interventions: Biological: Anti-Thymocyte Globulin - Rabbit; Biological: darTreg Infusion; Drug: Everolimus; Drug: Tacrolimus; Drug: Mycophenolate mofetil; Drug: Prednisone; Drug: Acetaminophen; Drug: Diphenhydramine; Drug: Anti-Infective Prophylaxis; Procedure: Leukapheresis; Procedure: Blood draws; Procedure: Liver biopsies; Procedure: Liver transplantation
- Cohort 3 - darTreg infusion,200 million(range100-240 million) (Experimental): At least 3 subjects will receive a single infusion dose of 200 million darTregs. Progression from one cohort to the next will depend on the cumulative incidence of sentinel adverse events.
  Interventions: Biological: Anti-Thymocyte Globulin - Rabbit; Biological: darTreg Infusion; Drug: Everolimus; Drug: Tacrolimus; Drug: Mycophenolate mofetil; Drug: Prednisone; Drug: Acetaminophen; Drug: Diphenhydramine; Drug: Anti-Infective Prophylaxis; Procedure: Leukapheresis; Procedure: Blood draws; Procedure: Liver biopsies; Procedure: Liver transplantation
- Cohort 4 - darTreg infusion,800 million(range 400-960 million) (Experimental): Six subjects will receive a single infusion of 800 million darTregs.
  Interventions: Biological: Anti-Thymocyte Globulin - Rabbit; Biological: darTreg Infusion; Drug: Everolimus; Drug: Tacrolimus; Drug: Mycophenolate mofetil; Drug: Prednisone; Drug: Acetaminophen; Drug: Diphenhydramine; Drug: Anti-Infective Prophylaxis; Procedure: Leukapheresis; Procedure: Blood draws; Procedure: Liver biopsies; Procedure: Liver transplantation

INTERVENTIONS:
Biological: Anti-Thymocyte Globulin - Rabbit — Liver transplantation/Treg-supportive immunosuppression (IS) treatment. Subjects will be given a dose range of 3.0-4.5 mg/kg total, in divided doses of 1.5 mg/kg/day. Subjects who meet eligibility criteria for Thymoglobulin® administration will be given 1.5 mg/kg intravenously (IV) on post-operative day 3, within 72 hours of transplantation. Additional doses of 1.5 mg/kg IV will be administered until CD3 count is <50/mm^3 or when the maximal dose of 4.5/mg/kg has been given.
  Other Names: ATG (Anti-Thymocyte Globulin); Thymoglobulin®
Biological: darTreg Infusion — A single dose darTreg infusion (Cohorts 2 - 4) will be received as per protocol.
  Other Names: Donor-Alloantigen-Reactive Regulatory T Cell Infusion
  Arms: Cohort 2 - darTreg infusion,50 million(range 25 to 60 million); Cohort 3 - darTreg infusion,200 million(range100-240 million); Cohort 4 - darTreg infusion,800 million(range 400-960 million)
Drug: Everolimus — Liver transplantation/Treg-supportive immunosuppression (IS) treatment. Subjects meeting eligibility criteria for Treg-supportive IS regimen will begin EVR no sooner than 30 days after liver transplantation and no later than 44 days after transplantation; with target trough levels of 6-8 μg/L.EVR target trough levels will be further reduced to 4-6 μg/L 24 - 26 weeks after transplantation.
  Other Names: EVR; Zortress®
Drug: Tacrolimus — Liver transplantation/Treg-supportive immunosuppression (IS) treatment. Between 30 and 44 days following transplant: Subjects who are not eliminated by Exclusion Criteria C1 (Protocol Section 14.3.1) will proceed in the study and receive either TAC-based or EVR- based IS, based on eligibility Criteria C2 (Section 4.3.4 )
  * TAC-based IS: reduce TAC trough level to 3-8 μg/dL; continue MMF
  * EVR-based IS: reduce TAC trough level to 3-8 μg/dL; EVR target trough level of 6-8 μg/dL; decrease then discontinue MMF
  Other Names: Prograf®
Drug: Mycophenolate mofetil — Liver transplantation/Treg-supportive immunosuppression (IS) treatment. 1000 mg total daily dose. MMF will be initiated within 24 hours of transplantation. MMF must be discontinued as soon as target EVR trough levels have been achieved.
  Other Names: MMF; Cellcept; Myfortic
Drug: Prednisone — Liver transplantation/Treg-supportive immunosuppression (IS) treatment. Solumedrol 500 mg will be given IV on the day of transplantation. Additional Solumedrol will be prescribed according to site-specific standard of care. Oral prednisone should be initiated once oral medication is tolerated.
  Other Names: Solumedrol
Drug: Acetaminophen — Pre-medication for single dose darTreg infusion (Cohorts 2 - 4). 650mg of acetaminophen will be administered intravenously or by mouth 30-60 minutes prior to the darTreg infusion.
  Other Names: Tylenol®
  Arms: Cohort 2 - darTreg infusion,50 million(range 25 to 60 million); Cohort 3 - darTreg infusion,200 million(range100-240 million); Cohort 4 - darTreg infusion,800 million(range 400-960 million)
Drug: Diphenhydramine — Pre-medication for single dose darTreg infusion (Cohorts 2 - 4). 25-50mg of diphenhydramine will be administered intravenously or by mouth 30-60 minutes prior to the darTreg infusion.
  Other Names: Diphenhydramine Hydrochloride
  Arms: Cohort 2 - darTreg infusion,50 million(range 25 to 60 million); Cohort 3 - darTreg infusion,200 million(range100-240 million); Cohort 4 - darTreg infusion,800 million(range 400-960 million)
Drug: Anti-Infective Prophylaxis — Intravenous ganciclovir and/or oral Valcyte will be administered for the prophylaxis of cytomegalovirus (CMV) and Epstein-Barr Virus (EBV) for at least six months after liver transplantation.
  Other Names: Antiviral Prophylaxis; ganciclovir; Cytovene; Valganciclovir; Valcyte
Procedure: Leukapheresis — Leukapheresis is necessary to ensure collection of adequate numbers of autologous Tregs to support ex vivo expansion of darTregs for infusion after liver transplantation.
  Participants enrolled in Cohorts 3 and 4 will undergo leukapheresis. Participants enrolled in Cohort 2 will have either whole blood collection or leukapheresis for the purpose of isolating autologous Tregs for later manufacture. If a cohort 2 subject has a hemoglobin level >/=10.5 gm/dL, he or she will undergo phlebotomy. If the patient has a hemoglobin level </=10.5 gm/dL and remains eligible for the study, the patient will undergo leukapheresis.
  Other Names: Leukocytapheresis
  Arms: Cohort 2 - darTreg infusion,50 million(range 25 to 60 million); Cohort 3 - darTreg infusion,200 million(range100-240 million); Cohort 4 - darTreg infusion,800 million(range 400-960 million)
Procedure: Blood draws — Blood draws are necessary to carefully and frequently evaluate allograft function after liver transplantation and treatment with Treg-supportive IS as well as after darTreg infusion. Peripheral blood samples will be collected and analyzed per protocol throughout subject participation in this study.
  Other Names: Venipuncture; Phlebotomy
Procedure: Liver biopsies — Subjects will have a liver biopsy for this study 12-14 weeks after transplantation. For subjects receiving darTregs, a second biopsy will be performed 7-10 days after darTregs infusion.
  Other Names: Liver biopsy samples
Procedure: Liver transplantation — Inclusion in this trial is in the setting of subjects defined as having end-stage liver disease and listed for primary solitary liver transplant.
  Other Names: Liver transplant

SUMMARY:
The purpose of this study is look at the safety of:

* Taking a specific combination of immunosuppressant drugs after liver transplantation
* Receiving one of three different doses of donor-alloantigen-reactive regulatory T cells (darTregs) while taking this specific combination of drugs

DETAILED DESCRIPTION:
After liver transplantation, immunosuppressants must be taken every day to prevent the body from injuring the transplanted liver by a process called rejection. People who take these drugs may experience side effects.

Studies show that some of body's cells, called T regulatory cells (Tregs), may play a part in accepting the transplanted liver. The investigators are learning about whether scientists can take Tregs from the blood of a liver transplant recipient and teach them to protect the transplanted liver from rejection. In the laboratory, the recipient Tregs are exposed to cells from the liver donor. Research data suggests that giving these "donor reactive" Tregs back to the transplant recipient might allow a liver transplant recipient to take lower doses of immunosuppressants, or perhaps to stop them altogether, without rejecting the liver.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who meet all of the following criteria are eligible for enrollment as study participants:

  * Able to understand and provide informed consent
  * End-stage liver disease and listed for primary solitary liver transplant
  * Have a calculated Model for End Stage Liver Disease (MELD) score ≤ 25 at the time of study entry/consent
  * Female and male subjects with reproductive potential must agree to use effective methods of birth control for the duration of the study.
  * If history of Hepatitis C Virus (HCV), have completed or are in current treatment for HCV AND have no detectable HCV RNA.
  * Subjects with HCC meeting Milan criteria.

Exclusion Criteria:

* Below are exclusion criteria to be assessed at study enrollment, prior to Stage 1 study procedures. Subjects who meet any of these criteria are not eligible for Stage 1 study procedures. Note that subjects in Cohort 1a or 1b will NOT undergo leukapheresis regardless of eligibility.

  * End stage liver disease secondary to autoimmune etiology (autoimmune hepatitis, primary biliary cirrhosis, or primary sclerosing cholangitis)
  * History of less than 5 years remission of malignancy, except for 1) HCC or 2) history of adequately treated in-situ cervical carcinoma, or adequately treated basal or squamous cell carcinoma of the skin.
  * History of previous organ, tissue or cell transplant
  * Serologic evidence of human immunodeficiency (HIV) 1 or -2 infection
  * Epstein-Barr Virus (EBV) or cytomegalovirus (CMV) sero-negativity (EBV or CMV naïve candidates)
  * Chronic use of systemic glucocorticoids or other Immunosuppression (IS), or biologic immunomodulators
  * Chronic condition requiring anti-coagulation after liver transplantation
  * Any chronic illness or prior treatment which, in the opinion of the investigator, precludes study participation
  * Participation in any other studies that involved investigational drugs or regimens in the preceding year
  * Received any vaccination within 28 days prior to leukapheresis or blood collection for Treg manufacture
  * Hemoglobin <9.0 g/dL within 10 days prior to screening
  * Neutrophils <1,500/μL within 10 days prior to screening
  * Platelets <40,000/μL within 10 days prior to screening
* Thymoglobulin Exclusion Criteria B (Stage 2):

  * Below are exclusion criteria to be assessed prior to administration of Thymoglobulin®. Subjects who meet any of these criteria should not receive Thymoglobulin®:

    * Calculated Model for End Stage Liver Disease (MELD) score >25 at the time of deceased donor liver transplant
    * Last alpha-fetoprotein (AFP) obtained prior to liver transplantation >400 μg/L for candidates with Hepatocellular Carcinoma (HCC)
    * Unacceptable Peripheral Blood Mononuclear Cells (PBMC) product for participants enrolled in Cohorts 2, 3, or 4 per the UCSF The Human Islet and Cellular Transplant Facility (HICTF) manufacturing specifications
    * Absence of donor spleen for any participants
    * Human leukocyte antigen (HLA)-DR (DR is one of class II antigens) matched to donor at both loci
    * Subject is < 21 or >70 years of age at the time of transplantation
    * Located in the intensive care unit 72 hours after transplantation
    * Hemoglobin <8.0 g/dL
    * Absolute neutrophil count <1,200/μL
    * Platelets <40,000/μL
    * Positive pregnancy test for females of child bearing potential
    * Unexpected histopathology on back table liver biopsy that contraindicates the initiation of Treg supportive IS regimen.
    * Development of a condition requiring chronic anti-coagulation.
    * Hypersensitivity to rabbit proteins or any excipient in Thymoglobulin®.
    * Detectable HCV RNA or less than six months after end of treatment for HCV at the time of transplantation (i.e., does not meet criteria for SVR).
  * Below are exclusion criteria to be assessed prior to conversion to Everolimus (EVR)-based IS regimen. (Assessed at day 30-44 after transplantation for continuation in the trial) All subjects regardless of eligibility for EVR conversion, with any of the following will not receive darTregs and will move into safety follow up:

    * Explanted liver with evidence of increased risk of recurrent cancer risk (hepatocellular (HCC) tumor burden exceeding the Milan criteria; presence of vascular invasion; cholangiocarcinoma morphology)
    * Insufficient depletion of recipient T cells, defined as a nadir CD3 count ≥50 cells μ/L (50 cells /mcL) or total lymphocyte count ≥ 0.1x 109/L if CD3 count is unavailable
    * Development of a condition requiring chronic anti-coagulation.
    * Clinical evidence of biliary obstruction
    * Alanine Aminotransferase (ALT) >2.0 x upper limit of normal (ULN)
    * Inability to taper off corticosteroids by 44 days (+/- 2 days) after transplant
    * Detectable circulating HCV RNA.

Everolimus Conversion Criteria C2 (assessed prior to conversion to EVR based IS regimen; EVR cannot be initiated prior to 30 days after liver transplantation). Subjects with any of the following will remain on TAC-based IS regimen.

* Evidence of hepatic artery stenosis or thrombosis by Doppler examination or angiography within 7 days prior to conversion
* Urine protein/creatinine ratio >1.0 within 7 days prior to conversion
* Calculated GFR less than 30 ml/min per MDRD4 (Modification of Diet in Renal Disease Study) equation within 7 days prior to conversion
* Physical examination documentation of abnormal wound healing or uncontrolled wound infection
* Hemoglobin <8.0 g/dL within 7 days prior to conversion
* Absolute neutrophil count <1,200/μL within 7 days prior to conversion
* Platelets <50,000/μL within 7 days prior to conversion

  *Below are exclusion criteria to be assessed prior to darTreg infusion for subjects in Cohorts 2, 3, and 4 only. Subjects in Cohort 2, 3, or 4 who meet any of these criteria should not receive a darTreg-infusion:
* Inability or unwillingness of participant to give additional written informed consent
* Unacceptable darTreg product
* Detectible circulating Epstein-Barr Virus (EBV) or cytomegalovirus (CMV) DNA within 10 days prior to darTreg infusion
* Detectible Hepatitis B Virus (HBV) DNA within 10 days prior to darTreg infusion
* Detectable circulating HCV RNA within 10 days prior to darTreg infusion.
* Alanine Aminotransferase (ALT) >1.5x upper limit of normal within 10 days of darTreg infusion
* Most recent, but not greater than 10 days prior to darTreg infusion,12 hour TAC trough levels of > 8 μg/L for all subjects
* Most recent, but not greater than 10 days prior to darTreg infusion,12 hour EVR trough levels of < 5 μg/L for subjects on EVR
* For subjects on EVR-based IS, received Mycophenolate Mofetil (MMF) within 10 days prior to darTreg infusion
* Evidence of acute rejection or chronic rejection according to Banff criteria on protocol allograft biopsy based on local assessment
* Received any vaccination within 14 days prior to darTreg infusion
* Positive pregnancy test for females of child bearing potential
* Inability or unwillingness of participant to comply with study protocol or procedures.
* Calculated glomerular filtration rate (eGFR) less than 40 ml/min per MDRD4 equation within 10 days prior to infusion.

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2014-12-17 (Actual); Primary Completion 2019-06-18 (Actual); Study Completion 2019-06-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sandy Feng, MD, PhD, Principal Investigator — University of California, San Francisco; Jeffrey Bluestone, PhD, Principal Investigator — University of California, San Francisco; Sang-Mo Kang, MD, FACS, Principal Investigator — University of California, San Francisco; Qizhi Tang, PhD, Principal Investigator — University of California, San Francisco
Locations (3):
- United States (3):
  - University of California, San Francisco, San Francisco, California
  - Northwestern University, Chicago, Illinois
  - Mayo Clinic, Rochester, Minnesota

REFERENCES:
- See also: National Institute of Allergy and Infectious Diseases (NIAID) website — https://www.niaid.nih.gov/

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1: Participants received Thymoglobulin®+EVR IS but will not receive darTregs
- Cohort 2: Participants received Thymoglobulin®+EVR IS and will receive a darTreg infusion of 50 million(range 25 to 60 million) cells.
- Cohort 3: Participants received Thymoglobulin®+EVR IS and will receive a darTreg infusion of 200 million(range 100 to 240 million) cells. No participants were enrolled in this cohort.
- Cohort 4: Participants received Thymoglobulin®+EVR IS and will receive a darTreg infusion of 800 million(range 400 to 960 million) cells. No participants were enrolled in this cohort.
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Started | 6 | 9 | 0 | 0
Completed | 6 | 8 | 0 | 0
Not Completed | 0 | 1 | 0 | 0
Not completed — Screen B Ineligible (Page 55, Protocol) | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants assigned to Treatment Cohorts after transplantation.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Total
Number analyzed (Participants) | 6 | 9 | 0 | 0 | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 5 | 6 | 0 | 0 | 11
  >=65 years | 1 | 3 | 0 | 0 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 59 (5.5) | 62 (4.2) |  |  | 61 (4.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 |  |  | 2
  Male | 4 | 9 |  |  | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 |  |  | 2
  Not Hispanic or Latino | 5 | 8 |  |  | 13
  Unknown or Not Reported | 0 | 0 |  |  | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 |  |  | 0
  Asian | 1 | 5 |  |  | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 |  |  | 0
  Black or African American | 0 | 0 |  |  | 0
  White | 5 | 4 |  |  | 9
  More than one race | 0 | 0 |  |  | 0
  Unknown or Not Reported | 0 | 0 |  |  | 0
Region of Enrollment [Number; unit: Count of Participants]
  United States | 6 | 9 |  |  | 15
Alanine Aminotransferase (ALT) [Mean (Standard Deviation); unit: U/L] — Normal Range in Adults: 7-41 U/L.
  U/L | 47.0 (66.6) | 216.4 (543.4) |  |  | 148.7 (421.5)
Alkaline Phosphatase [Mean (Standard Deviation); unit: U/L] — Normal Range in Adults: 33-96 U/L.
  U/L | 64.0 (17.3) | 102.8 (44.4) |  |  | 87.3 (40.2)
Gamma-Glutamyl Transferase (GGT) [Mean (Standard Deviation); unit: U/L] — Normal Range in Adults: 9-58 U/L.
  U/L | 40.0 (11.3) | 115.8 (97.0) |  |  | 100.6 (91.4)

OUTCOME MEASURES:

1. Primary Outcome: Percent of Participants With Biopsy-Proven Acute and/or Chronic Rejection
Description: Biopsy-proven acute rejection graded as Mild, Moderate or Severe, per 1997 Banff classification. Chronic Rejection graded using Banff 2000 classification.
  References: 1.) Banff Schema for Grading Liver Allograft Rejection: An International Consensus Document developed by an international panel of experts in liver transplantation pathology, hepatology, and surgery (Hepatology 1997; 25(3): 658-663). 2.) Update of the International Banff Schema for Liver Allograft Rejection: Working Recommendations for the Histopathologic Staging and Reporting of Chronic Rejection (Hepatology 2000; 31(3): 792-799).
Time Frame: Transplantation to 40 Weeks Post Transplantation
Population: All transplanted participants.
Measure: Number; unit: Percent of Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Number analyzed (Participants) | 6 | 9 | 0 | 0
Percent of Participants
  Mild Acute Rejection | 0 | 11.1 |  |
  Moderate Acute Rejection | 0 | 0 |  |
  Severe Acute Rejection | 0 | 0 |  |
  Chronic Rejection | 0 | 0 |  |

2. Primary Outcome: Percent of Participants With Grade 3 or Higher Infectious Adverse Event(s)
Description: The severity of infectious adverse events (AEs) was classified into grades as follows:
  * Grade 1 = asymptomatic; clinical or diagnostic observation only; intervention with oral antibiotic, antifungal, or antiviral agent only; no invasive intervention required
  * Grade 2 = symptomatic; intervention with intravenous antibiotic, antifungal, or antiviral agent; invasive intervention may be required
  * Grade 3 = any infection associated with hemodynamic compromise requiring pressors; any infection necessitating intensive care unit level of care; any infection necessitating operative intervention; any infection involving the central nervous system; any infection with a positive fungal blood culture; any proven or probable aspergillus infection; any tissue invasive fungal infection; any pneumocystis jiroveci infection
  * Grade 4 = life-threatening infection
  * Grade 5 = death resulting from infection
Time Frame: Transplantation to 40 Weeks Post Transplantation
Population: All transplanted participants.
Measure: Number; unit: Percent of Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Number analyzed (Participants) | 6 | 9 | 0 | 0
Percent of Participants | 0 | 11.1 |  |

3. Primary Outcome: Percent of Participants With Grade 3 or Higher Wound Complication(s) Adverse Event(s)
Description: The severity of adverse events (AEs) was classified into grades using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 4.0 (4/28/2009):
  * Grade 3 wound complications are defined as "Hernia without evidence of strangulation; fascial disruption/dehiscence; primary wound closure or revision by operative intervention indicated"
  * Grade 4 complications are defined as "Hernia with evidence of strangulation; major reconstruction flap, grafting, resection, or amputation indicated"
Time Frame: Transplantation to 40 Weeks Post Transplantation
Population: All transplanted participants.
Measure: Number; unit: Percent of Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Number analyzed (Participants) | 6 | 9 | 0 | 0
Percent of Participants | 0 | 0 |  |

4. Primary Outcome: Percent of Participants With Grade 2 or Higher Hematologic Adverse Events (AEs) of Anemia, Neutropenia, and/or Thrombocytopenia
Description: The severity of adverse events (AEs) was classified into grades using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 4.0 (4/28/2009):
  * Grade 1 = mild AE
  * Grade 2 = moderate AE
  * Grade 3 = severe and undesirable AE
  * Grade 4 = life-threatening or disabling AE
  * Grade 5 = death
Time Frame: Transplantation to 40 Weeks Post Transplantation
Population: All transplanted participants.
Measure: Number; unit: Percent of Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Number analyzed (Participants) | 6 | 9 | 0 | 0
Percent of Participants
  Anemia | 66.7 | 22.2 |  |
  Neutropenia | 16.7 | 0 |  |
  Thrombocytopenia | 16.7 | 0 |  |

5. Primary Outcome: Percent of Participants With Adverse Events (AEs) Attributable to the Donor Alloantigen Reactive Tregs (darTregs) Infusion
Description: AEs classified by the site investigator/clinician as possibly or definitely related to the study treatment, the Donor Alloantigen Reactive Tregs (darTregs) infusion. These AEs include:
  * infusion reaction
  * Grade 3 or higher cytokine release syndrome (Reference: National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 4.0 (4/28/2009) grading criteria
  * malignant cellular transformation.
Time Frame: Transplantation to 40 Weeks Post Transplantation
Population: Limited to participants that received darTreg infusion (N=1 study participant).
Measure: Number; unit: Percent of Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Number analyzed (Participants) | 0 | 1 | 0 | 0
Percent of Participants |  | 0 |  |

ADVERSE EVENTS:
Time Frame: 40 weeks
Groups:
- Cohort 1: Participants received Thymoglobulin® +EVR IS but will not receive darTregs
Arm/Group | Cohort 1 | Cohort 2
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/9
Serious Adverse Events (participants affected / at risk) | 4/6 | 4/9
Other Adverse Events (participants affected / at risk) | 6/6 | 6/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=6) | Cohort 2 (N=9)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0)
Oedema (General disorders) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 2 (2)
Biliary ischaemia (Hepatobiliary disorders) | 0 (0) | 0 (0)
Portal vein thrombosis (Hepatobiliary disorders) | 0 (0) | 0 (0)
Liver transplant rejection (Immune system disorders) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 1 (1) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Postoperative ileus (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0)
Failure to thrive (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0)
Calculus urinary (Renal and urinary disorders) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 1 (1) | 0 (0)
Hypocapnia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=6) | Cohort 2 (N=9)
Anaemia (Blood and lymphatic system disorders) | 4 (4) | 1 (1)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 1 (1) | 0 (0)
Oedema (General disorders) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0)
Biliary ischaemia (Hepatobiliary disorders) | 0 (0) | 1 (1)
Portal vein thrombosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Liver transplant rejection (Immune system disorders) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0)
Postoperative ileus (Injury, poisoning and procedural complications) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 2 (2) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 3 (3) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 0 (0) | 1 (1)
White blood cell count decreased (Investigations) | 1 (1) | 1 (1)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Calculus urinary (Renal and urinary disorders) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 0 (0)
Hypocapnia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Enrollment was terminated due to several factors:high number of ineligible subjects, slow enrollment, and manufacturing difficulties within the constraints of the funding period.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-08-01): https://cdn.clinicaltrials.gov/large-docs/19/NCT02188719/Prot_000.pdf
  • Statistical Analysis Plan (2020-05-06): https://cdn.clinicaltrials.gov/large-docs/19/NCT02188719/SAP_001.pdf